CLINICAL TRIAL: NCT04160559
Title: Green Tea Combined With Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer: A Randomized, Controlled Multicenter Clinical Study
Brief Title: Green Tea Combined With Chemotherapy in the Treatment of Advanced Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There are no suitable participants
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Clinical Professor, Xinqiao Hospital of Chongqing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-013
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer， green tea, chemotherapy，QOL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Control group: chemotherapy plus water, test group: chemotherapy plus green tea.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): chemotherapy plus water
  Interventions: Other: green tea
- Test group (Experimental): chemotherapy plus green tea
  Interventions: Other: green tea

INTERVENTIONS:
Other: green tea — The investigators require patients to regularly drink green tea during the trial period.

SUMMARY:
Patients with non-small cell lung cancer who met the inclusion and exclusion criteria were screened and randomly divided into control group and experimental group. Control group: chemotherapy plus water ,test group: chemotherapy plus green tea.

Primary endpoint: Assessment of changes in quality of life (QOL) after chemotherapy according to FACT-L (4th edition). A clinically significant change in the quality of life of lung cancer was defined as a FACT-L score change of ≥6 points from baseline, with <6 points defined as no clinically significant changes;

DETAILED DESCRIPTION:
Patients with non-small cell lung cancer who met the inclusion and exclusion criteria were screened and randomly divided into control group and experimental group. Control group: chemotherapy plus water (at least 3-5 cups per day, 100-120ml per cup), test group: chemotherapy plus green tea (patients drink tea from the beginning to the end of the test, patients drink moderately concentration of green tea 3-5 cups per day, 100-120ml per cup, and the monthly tea consumption is ≥100g. The tea concentration is defined that the amount of tea in the cup after boiling water is 50% or more which is "strong tea", 25% to 50% is "moderately concentrated tea", and less than 25% is "light tea"). The number of days of tea drinking by the patient is greater than or equal to 18 days per chemotherapy cycle.The quality of life of patients was assessed according to the Lung Cancer Quality of Life Scale (FACT-L (4th Edition)) and the Lung Cancer Symptom Scale (LCSS). Pre-chemotherapy quality of life scores were used as baseline. The evaluation was performed once before each chemotherapy, and the final quality of life assessment was performed within 1-4 weeks after the end of the fourth cycle of chemotherapy. A total of 5 quality of life assessments were completed. If the patient's condition progresses during chemotherapy, the assessment endpoint is when the disease progresses. Primary endpoint: Assessment of changes in quality of life (QOL) after chemotherapy according to FACT-L (4th edition). A clinically significant change in the quality of life of lung cancer was defined as a FACT-L score change of ≥6 points from baseline, with <6 points defined as no clinically significant changes;

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed NSCLC have evaluable lesions.
* ECOG PS：0-2分。
* Unintentional liver and kidney and other organic diseases, no other primary malignant tumors.
* Patients with clinical stage IIIB and IV who are scheduled for chemotherapy (first or second line).

Exclusion Criteria:

* Patients who have long-term tea drinking habits (more than 4 cups of green tea per day).
* Patients who have used immunological checkpoint inhibitors for more than 50%. Pregnant or lactating woman.
* The investigator judges other conditions that may affect the clinical research and the judgment of the research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-11 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL) according to FACT-L (4th edition). | 4-5 months
  A clinically significant change in the quality of life of lung cancer was defined as a FACT-L score change of ≥6 points from baseline, with <6 points defined as no clinically significant changes;

SECONDARY OUTCOMES:
Symptom changes assessed by the Lung Cancer Symptom Scale (LCSS). | 4-5 months
  A clinically significant change in symptoms was defined as a change in LCSS score from baseline ≥ 2 points, < 2 points defined as no clinically significant change.
Objective remission rate (ORR) . | 6 months
  Objective remission rate (ORR)
progression-free survival (PFS) | 6 months
  progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the second affiliated hospital of Army medical university, Chongqing, Chongqing Municipality
  - Xinqiao Hospital of Chongqing, Chongqing